CLINICAL TRIAL: NCT04106453
Title: Navigated Laparoscopic Microwave Ablation of Tumor Mimics in Pig Liver - an Ex-vivo Single Center Trial
Brief Title: Navigated Laparoscopic Microwave Ablation of Tumor Mimics in Pig Liver - an Ex-vivo Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Köln (Other)
Responsible Party: Principal Investigator, Roger Wahba, MD, PhD, Principal Investigator, Universitätsklinikum Köln
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 19-392
Record Dates: First submitted 2019-09-24; First posted 2019-09-27 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Liver Cancer; Surgery; Navigation, Spatial
Keywords: laparoscopy; navigation; microwave ablation; ultrasound guidance
MeSH Terms: conditions — Liver Neoplasms; Spatial Navigation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- navigated microwave ablation (Experimental): microwave ablation is performed laparoscopically with navigation
  Interventions: Procedure: navigated microwave ablation
- ultrasound guided microwave ablation (Active Comparator): microwave ablation is performed laparoscopically with ultrasound guidance
  Interventions: Procedure: ultrasound guided navigation

INTERVENTIONS:
Procedure: navigated microwave ablation — the laparoscopic microwave ablation in the pig liver is performed with the CasOne-Spot system
  Arms: navigated microwave ablation
Procedure: ultrasound guided navigation — the laparoscopic microwave ablation iin the pic liver is performed with ultrasound guidance
  Arms: ultrasound guided microwave ablation

SUMMARY:
In primary and secondary liver tumors microwave ablation could be an alternative to surgical resection.It could be performed laparoscopically. Under ultrasound control the microwave device is placed in the tumor.Therefore spatial orientation is challenging: the tumor is often missed and the failure rate is high. During learning curve this could lead to incomplete tumor ablation and high rate of local recurrence. Targeting systems could optimize that. The CasOne-SPOT-system is an innovative electromagnetic tracking and navigation system for laparoscopic microwave ablation. In this study targeting precision using the SPOT-System should be compared to conventional laparoscopic ultrasound-guided microwave ablation. Therefore tumor mimics (1-2cm) will be created in ex-vivo pig livers and microwave ablation will be performed ultrasound guided or ultrasound navigated. The ablation procedures will be performed by two novices and two experienced surgeons. Aim of this trial is to is to evaluate, if laparoscopic microwave ablation could be facilitated by the use of the SPOT-navigation system.

ELIGIBILITY:
Inclusion Criteria:

board certified surgeon with experienced liver surgery with/ without experience in laparoscopic microwave ablation

Exclusion Criteria:

* non

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-09-14 (Actual); Primary Completion 2020-01-14 (Actual); Study Completion 2020-02-04 (Actual)

PRIMARY OUTCOMES:
time to complete ablation | 0-10 minutes
  time from beginning of the targeting process until to complete ablation of the tumor mimic

SECONDARY OUTCOMES:
ablation completeness | up to 1 day
  the tumor in relation to the ablation figure is measures and the and and the completeness of the microwave ablation is evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Roger Wahba, MD, PhD, Principal Investigator — General, Visceral, Cancer and Transplant Surgery, University of Cologne
Locations (1):
- University of Cologne, Department of General, Visceral and Cancer Surgery, Cologne, Germany